CLINICAL TRIAL: NCT06524622
Title: Venous Excess Ultrasound Score (VExUS) Combined With Central Venous Pressure (CVP) to Predict Clinical Outcomes in Sepsis Participants
Brief Title: VExUS Combined With CVP to Predict Clinical Outcomes in Sepsis Participants
Status: Recruiting | Type: Observational
Sponsor: The Second People's Hospital of Yibin (Other)
Responsible Party: Principal Investigator, Wang Xueqian, Resident Physician, The Second People's Hospital of Yibin
Other Study IDs: SecondYibin
Record Dates: First submitted 2024-07-13; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Sepsis; Acute Kidney Injury
Keywords: VExUS; CVP; acute kidney injury; MAKE30; venous congestion
MeSH Terms: conditions — Sepsis; Acute Kidney Injury; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The ultrasound images of each participant

INTERVENTIONS:
Device: Point-of-care ultrasound (POCUS) — Point-of-care ultrasound (POCUS) measurements will be performed for all participants

SUMMARY:
Introduction:

Sepsis is a life-threatening organ dysfunction caused by a dysregulated host immune response to infection, and it is a common critical condition in the ICU. Early and timely fluid resuscitation is the cornerstone of sepsis treatment. However, excessive fluid loading can lead to interstitial edema and iatrogenic organ damage, particularly acute kidney injury (AKI). The VExUS grading system is a recently developed system that measures venous congestion through bedside ultrasound by assessing the blood flow waveforms of the portal vein, hepatic vein, and intrarenal veins, as well as the diameter of the inferior vena cava. Similarly, CVP is a commonly used indicator of venous congestion. The objective of this study is to Investigate the association between Venous Excess Ultrasound Score (VExUS), Central Venous Pressure (CVP) during the first three days of ICU admission, and the composite clinical outcome of major adverse kidney events within 30 days (MAKE 30) in sepsis participants.

Methods:

This study is a prospective, multicenter, observational study that will recruit at least 120 participants across multiple centers. Based on the definition of sepsis3.0, Participants with sepsis who are older than 18 years. Using Doppler ultrasound, Investigator will measure the IVC, HV, PV, and IRV, as well as lung ultrasound scores and cardiac-related parameters at 0-24 hours, 24-48 hours, and 48-72 hours after enrollment. Investigator will receive web-based educational courses, and image acquisition and interpretation will be adjudicated. The primary outcome is the relationship between VExUS score combined with CVP and MAKE 30 in sepsis participants.

DETAILED DESCRIPTION:
Study Title:

Association between VExUS Score Combined with CVP and Prediction of Clinical Outcomes in Septic participants: A Multicenter, Prospective, Observational Study.

Study Objective:

To investigate the relationship between VExUS score, CVP within the first 3 days of ICU admission in septic participants, and the composite clinical outcome of major kidney adverse events within 30 days (MAKE30).

Study Hypothesis:

The VExUS score and CVP in septic participants are related to the composite clinical outcome of major kidney adverse events within 30 days (MAKE 30), and the higher the VExUS score and CVP, the greater the risk of MAKE 30.

Outcome Measures:

Primary Outcome: Association between VExUS score, CVP, and MAKE30 in septic participants.

Secondary Outcomes: Incidence of AKI within 7 days and all-cause mortality within 30 days in septic participants.

Detailed Methods:

Case Selection:

participants admitted to the ICU of the participating research units between July, 2024 and ,January，2025 (the participating research units include: West China Hospital of Sichuan University, Sichuan Provincial People's Hospital, Mianyang Third People's Hospital, Affiliated Hospital of Southwest Medical University, Longquanyi District First People's Hospital, Pidu District People's Hospital, Wenjiang District People's Hospital, Xindu District Third People's Hospital,Yibin Second People's Hospital, etc.).

Data Collection:

After the participants were enrolled, participants demographic characteristics were collected: age, gender, height, weight, underlying comorbidities; main diagnosis upon ICU admission, site of infection, microbiological name, baseline serum creatinine level, etc. Collect data on diagnosing sepsis at Day1 (0-24hour), Day2 (24-48hour), Day3 (48-72hour), Day7, and Day30(Including Hemodynamic parameters, respiratory related indicators, neurologic related indicators, renal function indicators, cardiac markers, basic blood tests, infection indicators, severity scores, critical care ultrasound evaluation, Occurrence of AKI in day 7, AKI onset time, criteria, staging, Duration of mechanical ventilation, use of CRRT, vasopressor use, length of ICU stay, length of hospital stay, survival status, occurrence of MAKE30.)

Sample size calculation:

Preliminary calculation includes approximately 120 participants.

Statistical Analysis Methods:

Using SPSS software for statistical analysis. Normality test and homogeneity of variance test were conducted for quantitative data. Data that conform to normal distribution and homogeneity of variance are represented by mean ± standard deviation (x±s). Paired t-test is used for comparison between two groups, while one-way analysis of variance is used for comparison among multiple groups. For quantitative data that do not conform to normal distribution or homogeneity of variance, the median [interquartile range (IQR)] is used to represent the data, and non-parametric tests are used for comparison among multiple groups. Count data are expressed as frequency (percentage), and group comparisons are made using Fisher's exact probability test. Multiple logistic regression analysis is used to identify risk factors for AKI in sepsis participants. Receiver operating characteristic (ROC) curve analysis is conducted to assess the predictive value. Cox regression analysis is used to identify risk factors for mortality in sepsis AKI participants. P<0.05 indicates statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (age ≥ 18 years) with sepsis upon admission or during their stay in the ICU.

Exclusion Criteria:

* Age < 18 years
* Participants admitted to the ICU for < 24 hours
* Pregnant or lactating women
* Severe renal impairment (defined as baseline estimated glomerular filtration rate < 15 mL/min or requiring regular dialysis), including causes such as urinary tract obstruction, contrast agents, or nephrotoxic drugs
* Liver cirrhosis with portal hypertension
* Presence of urinary tract obstruction (which may affect IRVF waveform)
* Inability to resolve the primary disease
* Participants receiving palliative care
* Inability to obtain ultrasound images
* Inability to monitor CVP
* Refusal of monitoring by participants or their families

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the definition of sepsis3.0, Participants with sepsis who are older than 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes on MAKE30 | Day 30
  MAKE30 is : in-hospital mortality, receipt of new RRT, or persistent renal dysfunction defined as a final inpatient serum creatinine value ≥2 time baseline serum creatinine

SECONDARY OUTCOMES:
occurrence of AKI within 7 days | DAY 7
  Incidence of AKI from enrollment to 7 days post-enrollment
length of ICU stay and in-hospital stay | DAY30
  average length of ICU stay and in-hospital stay will be compared
VExUS score | DAY3
  difference of the VExUS score at day 1, 2, 3 day between groups.Higher score means more illness.
CVP value | DAY3
  difference of the CVP value at day 1, 2, 3 day between groups.Higher score means more illness.
All-cause mortality within 30 days | DAY30
  All-cause mortality within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: lianghai cao, Master's, Principal Investigator — Yibin Second People's Hospital, Associate Chief Physician
Locations (1):
- Point-of-care ultrasound (POCUS), Yibin, Sichuan, China

REFERENCES:
- [Result] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297
- [Result] Spiegel R, Teeter W, Sullivan S, Tupchong K, Mohammed N, Sutherland M, Leibner E, Rola P, Galvagno SM Jr, Murthi SB. The use of venous Doppler to predict adverse kidney events in a general ICU cohort. Crit Care. 2020 Oct 19;24(1):615. doi: 10.1186/s13054-020-03330-6. PMID 33076961